CLINICAL TRIAL: NCT06627946
Title: Ultrasound-guided Transversus Abdominis Plane Block Versus Local Wound Infiltration for Postoperative Analgesia After Cesarean Delivery: a Randomized Controlled Trial
Brief Title: Ultrasound-guided Transversus Abdominis Plane Block Versus Local Wound Infiltration (TAP_WI)
Acronym: TAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ministry of Health, Bhutan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 445; TAPStudy (Other: MoH)
Record Dates: First submitted 2024-09-20; First posted 2024-10-04 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2024-09

CONDITIONS: Transversus Abdominis Plane (TAP) Block; Wound Infiltration; Pain Score (VAS); Opioid Analgesia
Keywords: transversus abdominis plane block; Wound infiltration of local anesthesia; pain score; Opioid analgesia; cesarean section
MeSH Terms: conditions — Bites and Stings

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- TAP group (Experimental): Local anesthesia 0.25% bupivacine 20ml was administered at the transversus abdominis plane in TAP group (experiment)
  Interventions: Procedure: TAP group
- WI group (Active Comparator): Local anesthesia 0.25% bupivacine 20ml was administered or infiltrated along the cesarean wound in WI group as a an active comparator
  Interventions: Procedure: TAP group

INTERVENTIONS:
Procedure: TAP group — Local anesthesia 0.25% bupivacine was administered in the TAP plane

SUMMARY:
The goal of this clinical trial is to learn if transversus abdominis plane (TAP) block will reduce the cumulative opioid consumption compared to local wound infiltration (WI). It will also learn about the pain scores compared between TAP and WI groups. The main questions it aims to answer are:

Has the pain score after cesarean section been less in TAP compared to WI group? Has the cumulative consumption of opioids reduced in TAP as compared to WI group? Researchers will compare TAP group with WI group based on postoperative pain score and opioid used.

Participants will:

Be given intervention either TAP or WI during the cesarean section. Pain score will be recorded during the postoperative period at PACU, 6, 12 and 24 hours after cesarean section.

The postoperative pain will be rescued with opioid, and the cumulative use of opioids will be recorded.

DETAILED DESCRIPTION:
Study title:

Ultrasound-guided Transversus abdominis plane block versus local wound infiltration for postoperative analgesia after cesarean delivery: A randomized controlled trial

Study setting:

Bhutan is a small, landlocked country in the Himalayas, sandwiched between China and India. Its total population is over 0.7 million. 20 Healthcare in Bhutan is publicly owned and solely state-funded. It has a three-tiered health system with the primary health centers at the lowest level followed by district hospitals, regional referral hospitals, and the national referral hospital. 21 Jigme Dorji Wangchuk (JDW) National Referral Hospital is a tertiary referral hospital and a teaching hospital located in the capital city, Thimphu. The Department of Anesthesiology at JDW National Referral Hospital administers anesthesia in eight operation rooms. The department has nine anesthesiologists, eleven nurse anesthetists, seventeen anesthesia technicians, and five residents. The department also has pre-operative and post-anesthesia care unit (PACU) nurses.

In the pre-operative room, pregnant mothers posted for CS are received by the nurses, who complete preoperative documentation and administer prophylactic antibiotics. CS is performed by the resident under the supervision of a consultant or by a consultant obstetrician following a standard procedure under spinal anesthesia. Usually heavy bupivacaine ….mg (2.5ml) with fentanyl …mg (ml) is administered.

After the operation, patients are brought to PACU where the nurses monitor vitals and transfer them to postoperative wards once patients are awake and hemodynamically stable.

Study populations:

Women undergoing elective cesarean section in JDW National Referral Hospital

Inclusion criteria:

All elective cesarean sections performed under spinal anesthesia, with an American Society of Anesthesiologists physical status classification II (ASA II).

Exclusion criteria:

Those mothers underwent emergency cesarean section, contraindication to spinal anesthesia (increased intracranial pressure, coagulopathy, or local skin infection), hypersensitivity to any of the drugs used in the study, failed spinal anesthesia converted to general anesthesia, pre-existing pain syndromes, or with a history of recent opioid exposure, significant cardiovascular, renal, or hepatic disease, and fetal abnormalities or negative fetal outcomes were excluded from the study.

Study period:

The study was carried out from 1st January 2023 till 31st December 2023

Sample size:

The sample size was calculated using the G*Power version 3.1.97 with the following imputations- Test family: 't' tests; Statistical test: 'Mean' differences between two independent means (two groups); Type of power analysis: A priori, computer required sample size. Input parameters: two-tailed test, Type I error (α) = 0.05; Type II error (β) = 0.2; Power = 1-β = 0.8, allocation ratio N2/N1 = 1, and with an effect size (dz) 0.6. The total sample size (n) obtained was 90.

A drop-out rate of 10% was expected, and the total sample taken for the study was 100, divided equally into two groups TAP (n=50) and WI (n=50).

Study Procedure:

An ethical clearance was obtained from the Research Ethical Board of Health, Ministry of Health, Bhutan with Ref No: IRB/Approval/PN/2022-018/ 445, dated 10th November 2022.

All the pregnant mothers posted for elective CS were approached in the pre-operative room by the investigators and obtained written informed consent to participate in the study. Those mothers who voluntarily consented were recruited to the study after applying the inclusion criteria. Those mothers were briefed and familiarised with the visual analogue scale (VAS) for pain scores.

Randomization:

After recruitment, they were allocated into two groups, transversus abdominis plane (TAP) block and local wound infiltration (WI) consisting of 50 participants in each group. Allocation into two groups was done following a lottery system of randomization where each participant was made to pick up one from the basket containing 100 enclosed envelopes which consisted of 50 each for TAP and WI.

Blinding:

A single-blinded study was conducted where the study participants did not know which intervention they received.

In the operating room, patients were attached to anesthetic machines and monitored non-invasively for blood pressure, pulse rate, saturation, and electrocardiogram. All the patients were given intravenous crystalloid solution (Ringers Lactate) at a standard rate. Spinal anesthesia consisting of a preservative-free hyperbaric 0.5% bupivacaine of 1.8ml - 2.2ml was administered intrathecally at the L3 - L4 level using a 27G spinal needle. Failed spinal anesthesia and those converted to general anesthesia were excluded from the study.

After attaining an upper sensory level of T6 or higher, a standard CS with a Pfannenstiel incision was performed by the resident under supervision or by a consultant obstetrician. After the delivery of the baby, participants in both groups received oxytocin (30 units) through infusion and intravenous paracetamol (15mg/kg). Intraoperative complications were managed following the same protocol for both groups; bradycardia and hypotension were treated with inj ephedrine (….), and nausea/vomiting were managed inj metoclopramide (10mg).

Intervention:

In the TAP group, after completion of CS, the anesthesiologist performed a bilateral TAP block. The dividing screen was kept in place and the skin was cleaned with a 10% betadine solution. Under sterile precautions, using a linear ultrasound probe placed over the mid-axillary line at the midpoint between the costal margin and the iliac crest, the external oblique, internal oblique, and transversus abdominis muscles were identified. A 20 G nerve block needle was advanced under direct ultrasound vision through the skin, subcutaneous tissues, external oblique, and internal oblique, and once the needle tip reached the space between the internal oblique and the transversus abdominis muscle, a 20 ml of 0.25% bupivacaine was injected. A well-defined, hypoechoic, elliptical shape formation confirmed the correct site of injection. The same procedure was performed on the other side.

In Group WI, the local anesthetic wound infiltration was performed by the operating obstetrician. Before the skin closure, 20 ml of 0.25% bupivacaine was injected subcutaneously along the full length including both the upper and lower margins of the wound. The dividing screen was kept in place so the patient could not determine which pain intervention was being offered to them.

After the intervention following CS, participants were taken to the PACU and monitored for vitals. In the PACU, pain scores were assessed using the VAS by the investigators, and the postoperative complications including nausea, vomiting, pruritus, and the additional medications required in the PACU were recorded.

After they were shifted to the maternity ward, trained maternity nurses who were not a part of the study and unaware of the treatment modality, monitored and recorded the pain score, opioid consumption, and side effects at 6, 12, and 24 hours according to the questionnaire that was handed in the patient's file. Postoperative rescue analgesia was given according to the standard institute obstetricians protocol with scheduled oral paracetamol and intramuscular diclofenac sodium injections with on demand opioids (pethidine/tramadol/morphine). Ondansetron intravenous was offered for nausea and vomiting.

Study end-points:

Primary end-point was opioids consumption in the first 24hour after cesarean section.

Secondary end-point was VAS pain score (0-10) and side effects like post operative nausea, vomiting, sedation, and complications related to the procedure.

Data analysis:

Data were double-entered and validated using EpiData (version 3.1 for entry and version 2.2.2.183 for analysis, EpiData Association, Odense, Denmark). Data were exported and analyzed using SPSS (version 23). The Kolmogorov-Smirnov test was performed to test for the normality of the study data. Normally distributed continuous demographic and clinical characteristics variables were compared using student t-test. Non-normally distributed two independent variables were compared using Mann-Whitney test. The Chi square or Fisher's exact test was used to analyze categorical variables and presented in frequencies and percentages. The p-value of < 0.05 is considered statistically significant in the study.

ELIGIBILITY:
Inclusion Criteria:

1. All elective cesarean sections performed under spinal anesthesia,
2. American Society of Anesthesiologists physical status classification II (ASA II).

Exclusion Criteria:

1. Those mothers underwent emergency cesarean section
2. Contraindication to spinal anesthesia (increased intracranial pressure, coagulopathy, or local skin infection)
3. hypersensitivity to any of the drugs used in the study
4. Failed spinal anesthesia converted to general anesthesia
5. Pre-existing pain syndromes
6. History of recent opioid exposure
7. Significant cardiovascular, renal, or hepatic disease,
8. Fetal abnormalities or negative fetal outcomes were excluded from the study

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Pregnant women
Enrollment: 100 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
To compare cumulative consumption of opioids in the first 24 hours after cesarean section | within 24 hours postoperative period
  Cumulative use of Inj. morphine during the postoperative period was significantly less in the TAP group than in the WI group (5.4 ± 0.9 Vs 6.1 ± 0.6, p=0.017)

SECONDARY OUTCOMES:
To compare the pain score using the Visual Analogue Scale between the intervention (TAP) and comparator (WI) group | within 6, 12 and 24 hours postoperative period
  The postoperative pain score was significantly lower in the intervention (TAP) group where patients received ultrasound-guided transversus abdominis plane block as compared to a comparative (WI) group who received wound infiltration of local anesthesia (0.62 ± 0.87 Vs 1.22 ± 1.44 respectively, p-value 0.013) at the post-anesthesia care unit (PACU).
To compare the postoperative complications between the intervention (TAP) group with the comparator (WI) group. | Within first 24 hours postoperative period
  Postoperative complications were reported in over 15% (15/99) of the patients. Postoperative complications reported were less in the experimental (TAP) group as compared to the WI group.

CONTACTS AND LOCATIONS:
Overall Officials: Yeshey Dorjey, MD, Principal Investigator — Phuentsholing General Hospital
Locations (1):
- Yeshey Dorjey, Phuentsholing, Phuentsholing, Chukha, Bhutan

IPD SHARING:
Plan to Share IPD: No